CLINICAL TRIAL: NCT01598961
Title: Determination of Target of Adequate Partial Neuromuscular Blockade for Electrophysiologic Monitoring During Microvascular Decompression Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Jin Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2012-03-089-001
Record Dates: First submitted 2012-05-12; First posted 2012-05-15 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Hemifacial Spasm; Microvascular Decompression; Lateral Spread Response Monitoring
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TOF count-guided group (Active Comparator): Using partial neuromuscular blockade to maintain train-of-four response of two, TOF response measured by the neuromuscular transmission module (NMT module)
  Interventions: Other: TOF count-guided partial NMB
- T1/Tc amplitude group (Active Comparator): Using partial neuromuscular blockade to maintain T1/Tc amplitude of 50%, T1/Tc amplitude measured by the neuromuscular transmission module (NMT)
  Interventions: Other: T1/Tc guided partial NMB
- No neuromuscular blockade group (Experimental): to maintain no neuromuscular blockade during LSR monitoring except the intubation dose during anesthetic induction
  Interventions: Other: No NMB

INTERVENTIONS:
Other: TOF count-guided partial NMB — Using partial neuromuscular blockade to maintain train-of-four response of two, TOF response measured by the neuromuscular transmission module (NMT module)
  Arms: TOF count-guided group
Other: T1/Tc guided partial NMB — Using partial neuromuscular blockade to maintain T1/Tc amplitude of 50%, T1/Tc amplitude measured by the neuromuscular transmission module (NMT)
  Arms: T1/Tc amplitude group
Other: No NMB — to maintain no neuromuscular blockade during LSR monitoring except the intubation dose during anesthetic induction
  Arms: No neuromuscular blockade group

SUMMARY:
There have been reports of monitoring LSR during MVD surgery helps predicting the clinical outcome of MVD.However, there have been no evidence of which degree of partial neuromuscular blockade should be performed or no neuromuscular blockade could be performed during LSR monitoring. Therefore, we performed a randomized controlled trial to evaluate the effect of different degree of partial neuromuscular blockade, including no neuromuscular blockade on the LSR monitoring for MVD surgery.

DETAILED DESCRIPTION:
Hemifacial spasm develops by vascular compression of facial nerve at the root exit zone from brain stem. Microvascular decompression (MVD) is known for its curative treatment. Lateral spread response (LSR) is a kind of pathologic electromyographic (EMG) wave form which develops when facial nerve is compressed by vessel. There have been reports of monitoring LSR during MVD surgery helps predicting the clinical outcome of MVD.

As neuromuscular blockade during LSR monitoring decreases the amplitude of EMG, partial neuromuscular blockade is usually maintained during general anesthesia for MVD. However, there have been no evidence of which degree of partial neuromuscular blockade should be performed or no neuromuscular blockade could be performed during LSR monitoring. Therefore, we performed a randomized controlled trial to evaluate the effect of different degree of partial neuromuscular blockade, including no neuromuscular blockade on the LSR monitoring for MVD surgery.

ELIGIBILITY:
Inclusion Criteria:

* Those who undergo microvascular decompression by diagnosis of hemifacial spasm in our institution

Exclusion Criteria:

* Patients were excluded from the study if they had any of following: severe cardiopulmonary disorder with hemodynamic unstability (pulmonary hypertension, cardiomyopathy, mechanical ventilation, American Society of Anesthesiologists physical status III or more), severe hepatic or renal disease.
* Those who can not undergo MEP monitoring due to central or peripheral neuromuscular disease, e.g. cerebral palsy, myasthenia gravis, acute spinal injury, neurologic shock

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Lateral spread response | baseline (30 min after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist at baseline (30 min after anesthetic induction)
Lateral spread response | before dura opening (45 minute after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist before dura opening
Lateral spread response | after dura opening (60 min after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist after dura opening (one hour after anesthetic induction)
Lateral spread response | before facial nerve decompression (90 minutes after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist before facial nerve decompression (90 minutes after anesthetic induction)
Lateral spread response | after facial nerve decompression (120 min after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist after facial nerve decompression (2 hour after anesthetic induction)
Lateral spread response | after dura closure (150 min after anesthetic induction)
  Lateral spread response of electromyography measured by electrophysiologist after dura closure (150 min after anesthetic induction)

SECONDARY OUTCOMES:
Train-of-four response | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  Train-of-four response to ulnar nerve electrical stimulation measured by NMT module at six time-points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
T1/Tc amplitude | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  T1/Tc amplitude as a reponse to ulnar nerve stimulation measured by NMT module at six time points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
incidence of patients' spontaneous movements or respiration | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  incidence of patients' spontaneous movements or respiration measured by anesthesiologists or reported by surgeon at six time points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
Mean blood pressure (mmHg) | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  mean blood pressure measured by anesthesiologists at six time points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
heart rate (beats/min) | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  heart rate measured by anesthesiologists at six time points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
pulse oximetry (oxygen saturation, %) | Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)
  pulse oximetry measured by anesthesiologists at six time points; Baseline (30min), Before dura open (45 min), After dura open (60 min), Before decompression (90 min), After decompression (120 min), After dura close (150 min after anesthetic induction)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Jin Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, South Korea